CLINICAL TRIAL: NCT00381121
Title: Michigan Nephrology Research BioBank for Molecular Analysis of Renal Disease "Nephrology Research BioBank"
Brief Title: University of Michigan "Nephrology Research BioBank"
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Matthias Kretzler, Professor of Medicine, University of Michigan
Other Study IDs: HUM 4729
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease
Keywords: Tissue Biobank; molecular markers; molecular pathways
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, urine
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Kidney disease cohort: Individuals with a clinically indicated biopsy are recruited and/or surplus tissue that remains from past clinical interventions is obtained.

SUMMARY:
The purpose of the study is to create a Nephrology Tissue Biobank enabling the study of kidney disease from the perspectives of epidemiology, genetics and molecular biology.

DETAILED DESCRIPTION:
Each year chronic kidney disease (CKD) claims the lives of millions of people worldwide. Costs for patient care are in excess of 2.4 billion dollars in the US alone. At the moment most kidney diseases are of unknown etiology, are classified according to a microscopic description of the kidney tissue obtained on biopsy and are treated with non-specific therapies.

Each kidney contains millions of filter units called nephrons. The nephron consists of a glomerulus and a tubule. The glomerulus filters the blood of waste products, while retaining larger molecules that are required for the body to function properly. The filtered fluid then passes through the tubule, where salts, acids and water are regulated to keep the body in a normal metabolic state. After the filtered fluid passes through the tubule it is collected in the bladder as urine. Diseases, which affect the glomeruli or tubules result in kidney damage. Once kidney function is lost it is generally not recoverable and the only option for a patient's survival is dialysis or transplantation.

The purpose of this study is to provide a platform, which will enable researchers with different areas of expertise, to investigate the molecular markers and pathways of kidney disease and its progression. Our goal is to increase our understanding of kidney health issues and to develop new prevention and treatment strategies which will be shared with the medical community and the public.

Study description:

Individuals seen in the nephrology clinic at the University of Michigan will be eligible to enroll in this study. Their clinical data will be recorded, blood and urine samples will be collected and if a biopsy is performed as a part of their standard medical care then a small sample will be reserved for use in the study after all pathological evaluations required for patient care are completed. Biological samples will be available for biochemical, molecular biological and genetic testing and for correlation of these parameters to the individuals clinical data in future studies.

Significance:

Advances in the understanding of kidney disease may 1) provide methods of early detection of disease, 2) identify molecular markers that will help physician prescribe the most appropriate and beneficial treatments, 3) identify targets for the development of new treatments, and 4) decrease the enormous cost of caring for individuals with CKD.

Aim:

1. Create a biobank enabling the study of kidney disease from the perspectives of epidemiology, genetics and molecular biology.
2. Create a resource for the study of kidney disease, which will enable the researchers at the University of Michigan to work collaboratively toward the elucidation of the molecular pathways, which cause kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Men, women and children undergoing kidney and/or pancreas biopsy at the University of Michigan

Exclusion Criteria:

* Individuals not willing to provide consent (for prospective biopsy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Renal disease patients undergoing diagnostic workup
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2006-09; Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kretzler,, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Schmid H, Henger A, Kretzler M. Molecular approaches to chronic kidney disease. Curr Opin Nephrol Hypertens. 2006 Mar;15(2):123-9. doi: 10.1097/01.mnh.0000214770.11609.fb. PMID 16481877